CLINICAL TRIAL: NCT04117477
Title: Healthcare Associated Infection Reduction in Stem Cell Transplant Patients: a Randomized, Double-blind, Placebo-controlled Study Evaluating Twice Daily Xylitol Administration
Brief Title: Xylitol - Healthcare Associated Infection Reduction in Stem Cell Transplant Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: A new multisite study was opened in place of this study.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-0261
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Allogeneic Hematopoietic Cell Transplantation
MeSH Terms: interventions — Xylitol

STUDY DESIGN:
Intervention Model Description: 1:1, randomized, double-blind, placebo-controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Xylitol wipes (Experimental)
  Interventions: Drug: Xylitol
- Placebo wipes (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Xylitol — Xylitol dental wipes
  Arms: Xylitol wipes
Other: Placebo — Placebo dental wipes
  Arms: Placebo wipes

SUMMARY:
The central hypothesis is that daily dental xylitol wipes, in addition to current oral care practice, are effective at reducing BSI from oral organisms, and decreasing the incidence of gingivitis, oral plaque, and oral ulcerations after SCT.

DETAILED DESCRIPTION:
Our long-term goal is to develop and disseminate clinically relevant, and easily adoptable strategies to prevent BSI and improve outcomes after SCT. The overall objective of this proposal is to identify a clinically effective strategy to prevent or reduce BSI secondary to bacterial translocation through oral injured mucosa .

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age undergoing SCT.

Exclusion Criteria:

* Prior proton or photon radiation treatment for cancer of the oral cavity, head or neck; cranial boost in patients receiving total body irradiation; known history of allergy to xylitol; inability to use a mouth rinse or dental wipes.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Incidence of bacteremia in the first 30 days post-HSCT with oral organisms | 30 days
Incidence of bacteremia in the first 30 days post-HSCT with any organism | 30 days

SECONDARY OUTCOMES:
Incidence of dental plaque | 30 days
Incidence of gingival inflammation | 30 days
Incidence of mucosal ulceration | 30 days
Incidence of oral mucositis | 30 days
Incidence of oral microbiome diversity | 30 days
Incidence of oral pathogenic bacteria burden | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States